CLINICAL TRIAL: NCT04285762
Title: Supermicrosurgical Lymphatic Venous Anastomosis for Lymphedema Treatment
Brief Title: Supermicrosurgical LVA for Lymphedema Treatment
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201801774B0
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent supermicrosurgical LVA: Patients underwent supermicrosurgical LVA by a single surgeon from March 2016 to October 2018.
  Interventions: Other: LVEEA; Other: LVESA; Other: LVSEA

INTERVENTIONS:
Other: LVEEA — lymphaticovenous end-to-end
Other: LVESA — lymphaticovenous end-to-side
Other: LVSEA — lymphaticovenous side-to-end

SUMMARY:
LVA orientations such as lymphaticovenous end-to-end (LVEEA), end-to-side (LVESA), and side-to-end (LVSEA) are commonly performed. Each orientation has its own advantages and disadvantages. The key factors affecting the type of anastomotic orientation are the sizes of the LVs and the RVs, and the relative distance between them. Most published literatures have focused on LVSEA2-9, which is considered to be the most efficient. With one anastomosis in LVSEA, the RV is able to drain both the antegrade and retrograde lymphatic flow. Nevertheless, how to determine the anastomotic orientation has remained ambiguous. In this study, we aimed to establish the basis of selecting the proper anastomotic orientation, based on the size and comparative size discrepancy between LV and RV. To the best of our knowledge, this is the first report to focus on this subject.

ELIGIBILITY:
Inclusion Criteria:

* lymphedematous lower limbs (International Society of Lymphology stage I-III) between March 2016 to October 2018 were included

Exclusion Criteria:

* Patients whose data were missing will be excluded.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective observational study was approved by the institutional review board in our hospital. From March 2016 to October 2018, 100 patients with 103 lymphedematous lower limbs (International Society of Lymphology stage I-III) were included. All the patients underwent supermicrosurgical LVA performed by a single surgeon using a high-power microscope.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
survival or failure | up to 3 months
  The primary free flap outcome was determined as its survival or failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan